CLINICAL TRIAL: NCT07404267
Title: The Utility of Oxygen Reserve Index Guidance in Inspiratory Oxygen Titration for Patients Undergoing Surgery in the Beach Chair Position: A Prospective Comparative Study
Brief Title: Oxygen Reserve Index-Guided Oxygen Titration During Surgery in the Beach Chair Position
Acronym: ORI-BCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Çağla Sancak, Resident in Anesthesiology, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORI-FIO2-BCP-2025; 2025/234 (Other: Sancaktepe Şehit Prof. Dr. İlhan Varank education and research hospital Ethics Committee Approval Number)
Record Dates: First submitted 2026-01-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Hyperoxemia; Intraoperative Oxygen Therapy; Beach Chair Position; Cerebral Oxygenation
Keywords: Oxygen Reserve Index; ORİ; FiO2 titration; Hyperoxia; Pulse oximetry; Arterial blood gas; Near-infrared spectroscopy; General anesthesia; Beach chair position; Orthopedic surgery
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups in which inspiratory oxygen fraction (FiO₂) is titrated either using combined Oxygen Reserve Index (ORi) and SpO₂ guidance or SpO₂ guidance alone throughout surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORi-Guided FiO₂ Titration (Experimental): Inspiratory oxygen fraction (FiO₂) will be titrated using combined Oxygen Reserve Index (ORi) and peripheral oxygen saturation (SpO₂) monitoring throughout surgery.
  Interventions: Other: ORi-Guided FiO₂ Titration
- SpO₂-Guided Oxygen Titration (Active Comparator): Inspiratory oxygen fraction (FiO₂) will be titrated based on peripheral oxygen saturation (SpO₂) values according to routine clinical practice.
  Interventions: Other: SpO₂-Guided FiO₂ Titration

INTERVENTIONS:
Other: ORi-Guided FiO₂ Titration — Inspiratory oxygen fraction (FiO₂) will be adjusted throughout surgery using combined Oxygen Reserve Index (ORi) and peripheral oxygen saturation (SpO₂) monitoring. FiO₂ will be titrated to maintain ORi values between 0.2 and 0.5, with reassessment every 2-3 minutes.
  Arms: ORi-Guided FiO₂ Titration
Other: SpO₂-Guided FiO₂ Titration — FiO₂ will be adjusted to maintain SpO₂ at or above 98% throughout surgery.
  Arms: SpO₂-Guided Oxygen Titration

SUMMARY:
This study aims to evaluate whether guidance by the Oxygen Reserve Index (ORi) improves inspiratory oxygen fraction (FiO₂) titration compared with conventional pulse oximetry (SpO₂)-guided oxygen administration in adult patients undergoing surgery in the beach chair position.

Oxygen therapy is routinely used during general anesthesia to prevent hypoxemia; however, excessive oxygen administration may result in hyperoxia, which has been associated with adverse cardiovascular and pulmonary effects. Standard pulse oximetry may not adequately detect hyperoxia when oxygen saturation values are high.

In this prospective comparative study, patients will receive oxygen titration guided either by SpO₂ alone or by combined ORi and SpO₂ monitoring. The primary outcome is the incidence of intraoperative hyperoxemia, assessed by arterial blood gas analysis. Secondary outcomes include intraoperative oxygenation parameters and hemodynamic variables.

DETAILED DESCRIPTION:
This prospective study will be conducted in adult patients (ASA physical status I-III) undergoing elective orthopedic surgery in the beach chair position under general anesthesia. Following approval by the institutional ethics committee and acquisition of written informed consent, eligible patients will be included in the study.

Standard monitoring will include electrocardiography, noninvasive blood pressure, peripheral oxygen saturation (SpO₂), bispectral index (BIS), perfusion index (PI), pleth variability index (PVI), near-infrared spectroscopy (NIRS), and multiwavelength pulse co-oximetry for Oxygen Reserve Index (ORi) monitoring. Invasive arterial blood pressure monitoring will be established via radial arterial cannulation to allow continuous hemodynamic monitoring and arterial blood gas sampling.

General anesthesia will be induced with intravenous propofol, fentanyl, and rocuronium, followed by orotracheal intubation. Mechanical ventilation will be applied in volume-controlled mode with lung-protective settings. Anesthesia will be maintained using sevoflurane and remifentanil infusion, targeting bispectral index values between 40 and 60.

From anesthesia induction onward, inspiratory oxygen fraction (FiO₂) will be titrated either according to SpO₂ values alone or using combined ORi and SpO₂ guidance. In the ORi-guided group, FiO₂ adjustments will aim to maintain ORi values between 0.2 and 0.5, with reassessment at regular intervals. In the SpO₂-guided group, FiO₂ will be adjusted to maintain SpO₂ values at or above 98%, in accordance with routine clinical practice.

Hemodynamic parameters, oxygenation variables, ORi values, and cerebral oxygenation assessed by NIRS will be recorded at predefined time points during surgery and recovery. Arterial blood gas analysis will be performed to determine PaO₂ and arterial oxygen saturation.

Hyperoxemia will be defined as a PaO₂ value of 100 mmHg or greater and classified as mild or severe. The primary outcome of the study is the incidence of intraoperative severe hyperoxemia. Secondary outcomes include overall oxygenation profiles and intraoperative hemodynamic stability.

The results of this study are expected to provide evidence regarding the utility of ORi-guided oxygen titration in reducing unnecessary hyperoxia during surgery performed in the beach chair position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 65 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective orthopedic surgery in the beach chair position
* Body mass index (BMI) <35 kg/m²
* Ability to provide written informed consent

Exclusion Criteria:

* Age <18 or ≥65 years
* Finger deformities preventing the use of Oxygen Reserve Index (ORi) monitoring
* Severe anemia (hemoglobin <8 g/dL)
* Pregnancy
* Refusal or inability to provide informed consent
* History of stroke or significant vascular pathology
* Severe cardiac or respiratory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intraoperative Severe Hyperoxemia | Perioperative/Periprocedural
  Severe hyperoxemia will be defined as an arterial partial pressure of oxygen (PaO2) ≥200 mmHg, measured by arterial blood gas analysis at predefined intraoperative time points.

SECONDARY OUTCOMES:
Mean Peripheral Oxygen Saturation (SpO2) During Surgery | Perioperative/Periprocedural
  Peripheral oxygen saturation (SpO2) measured continuously during surgery using standard pulse oximetry.
Mean Oxygen Reserve Index (ORi) During Surgery | Perioperative/Periprocedural
  Oxygen Reserve Index (ORi) values recorded intraoperatively to evaluate oxygenation status.
Mean Fraction of Inspired Oxygen (FiO₂) During Surgery | Perioperative/Periprocedural
  Mean fraction of inspired oxygen (FiO₂) expressed as percentage (%), averaged over the surgical period.
Mean Cerebral Oxygen Saturation Measured by Near-Infrared Spectroscopy During Surgery | Intraoperative period (from induction of anesthesia to end of surgery)
  Cerebral regional oxygen saturation values measured intraoperatively using near-infrared spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: cagla sancak, MD, Principal Investigator — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Istanbul Provincial Health Directorate Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)